CLINICAL TRIAL: NCT01363362
Title: Effect of Selective Lasertrabeculoplasty (SLT) on Ocular Hemodynamics in Glaucoma
Brief Title: Selective Lasertrabeculoplasty and Ocular Hemodynamics in Glaucoma
Acronym: SLT/OBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Principal Investigator, Technische Universität Dresden
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLT/OBF_EK 398122010
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Glaucoma
Keywords: Selective Laser Trabeculoplasty; pulsatile ocular blood flow
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- glaucoma patients (Experimental): Glaucoma patients undergoing selective laser trabeculoplasty for further IOP reduction
  Interventions: Procedure: Selective Laser Trabeculoplasty

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — 360° selective laser trabeculoplasty, 100 non-overlapping spots, energy 0,5-1,2 mJ
  Other Names: Lasertrabeculoplasty

SUMMARY:
Selective Laser Trabeculoplasty (SLT) is known to reduce intraocular pressure in glaucoma patients. This study investigates, if there are changes in different ocular hemodynamic parameters prior and after SLT.

DETAILED DESCRIPTION:
Ocular blood flow, ocular pulse amplitude and ocular pulse volume are measured with the Blood Flow Analyzer (Paradigm Medical Industries, Inc.) prior and 3 month after SLT.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patient
* over 18 years
* needs further intraocular pressure regulation

Exclusion Criteria:

* age under 18 years
* debilitated
* no glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in ocular hemodynamics after Selective Laser Trabeculoplasty (SLT) | baseline and 3 month
  Pulsatile ocular blood flow, ocular pulse amplitude and ocular pulse volume are measured prior and 3 month after SLT with the Blood Flow Analyzer (Paradigm Medical Industries, Inc.)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz E Pillunat, Prof. MD, Study Chair — University Eye Clinic Dresden
Locations (1):
- University Eye Clinic Dresden, Dresden, Saxony, Germany